CLINICAL TRIAL: NCT00535314
Title: A Multicenter, Phase II, Randomized, Open Label Trial of 2 Dose Levels of RTA 402 in Patients With Advanced Malignant Melanoma
Brief Title: Study of Two Dose Levels of RTA 402 in Patients With Advanced Malignant Melanoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTA 402-C-0704
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Malignant Melanoma
Keywords: Melanoma
MeSH Terms: conditions — Melanoma | interventions — ORF 50 transactivator

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RTA 402 Dose1 (Experimental): Dose1 of RTA 402 to be administered orally once daily for 28 consecutive days, for up to 18 months.
  Interventions: Drug: RTA 402 Dose1
- RTA 402 Dose2 (Experimental): Dose2 of RTA 402 to be administered orally once daily for 28 consecutive days, for up to 18 months.
  Interventions: Drug: RTA 402 Dose2

INTERVENTIONS:
Drug: RTA 402 Dose1
  Arms: RTA 402 Dose1
Drug: RTA 402 Dose2
  Arms: RTA 402 Dose2

SUMMARY:
The primary purpose of the study is to determine the proportion of patients without progression at 6-months in patients with unresectable Stage III or Stage IV melanoma who are taking RTA 402.

DETAILED DESCRIPTION:
This is a phase II, open label, randomized study in patients with unresectable Stage III or Stage IV malignant melanoma. Patients will be randomly assigned to two different doses of RTA 402 administered orally once daily for 28 consecutive days, for up to 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 18 years of age
* Confirmed diagnosis of malignant (unresectable Stage III or Stage IV) melanoma
* Measurable disease, defined as at least 1 lesion which measures more than or equal to 20 mm by conventional techniques, or more than or equal to 10 mm by spiral CT scan, or cutaneous lesion of greater than or equal to 10 mm by caliper.
* May have received no more than 1 prior chemotherapy for metastatic disease.
* May have received prior vaccine therapy in the adjuvant setting.
* May have received cytokine therapy in the adjuvant setting and/or 1 prior cytokine therapy for metastatic disease.
* ECOG performance of 0-1
* Must have adequate liver and renal function documented by laboratory test results.
* Must have adequate bone marrow function documented by lab results.
* Must have completed any prior chemotherapy, immunotherapy, radiation, biological, or other investigational cancer therapy at least 4 weeks prior to starting this study, and have recovered from all acute side effects. Patients receiving mitomycin C or nitrosoureas must be 6 weeks from the last administration of chemotherapy.
* Man or woman must agree to practice effective contraception during the study and for at least 2 months after the last dose of RTA 402.
* Must have life expectancy of more than 3 months.
* Must be willing and able to sign the informed consent form.
* Must be willing and able to take and document oral doses of RTA 402.

Exclusion Criteria:

* May have received no more than 1 prior chemotherapy.
* May have received no more than 1 prior cytokine therapy for metastatic disease.
* Diagnosis of ocular melanoma.
* Inability to swallow tablets or capsules
* Symptomatic malabsorptive disorder (eg, Crohn's Disease), or removal of either the terminal ileus or more than 2/3 of the small intestine.
* Active brain metastases or primary central nervous system malignancies; patients with a previously treated brain metastasis may be included provided that there is no requirement for steroids and no evidence for progression for greater than or equal to 8 weeks after treatment.
* Active second malignancy.
* Weight loss greater than or equal to 10% over the 6 weeks prior to dosing
* Pregnant or breast feeding
* Clinically significant illnesses which could compromise participation in the study, including: uncontrolled diabetes; active or uncontrolled infection; acute or chronic liver disease; confirmed diagnosis of HIV infection; uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction within the last 6 months, or uncontrolled cardiac arrhythmia.
* Psychiatric illness that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
To determine the proportion of patients without progression at 6 months in patients with unresectable Stage III or Stage IV melanoma treated with RTA 402.

SECONDARY OUTCOMES:
To determine the overall response rate and duration of responses

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/